CLINICAL TRIAL: NCT01870375
Title: Longitudinal Studies of Brain Structure and Function in MPS Disorders
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Lysosomal Disease Network (Other)
Responsible Party: Sponsor
Other Study IDs: 0905M65804; U54NS065768 (NIH); 0905M65804 (Other: Univ. of Minnesota IRB Identifier Number)
Record Dates: First submitted 2011-08-02; First posted 2013-06-06 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Mucopolysaccharidosis Type I; Mucopolysaccharidosis Type II; Mucopolysaccharidosis Type VI; Mucopolysaccharidosis Type IV; Mucopolysaccharidosis Type VII
Keywords: Mucopolysaccharidosis; Longitudinal; Brain; Cognition; Quality-of-Life; Hurler syndrome; Hunter syndrome; Hurler-Scheie syndrome; Scheie syndrome; Maroteaux-Lamy syndrome; MPS I; MPS II; MPS VI; Mucopolysaccharidosis type I; Mucopolysaccharidosis type II; Mucopolysaccharidosis type VI; MPS IV; MPS VII; Mucopolysaccharidosis type IV; Mucopolysaccharidosis type VII; Morquio syndrome; Sly syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI; Mucopolysaccharidosis IV; Mucopolysaccharidosis VII; Mucopolysaccharidoses; Sudden Infant Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- MPS IH, MPS IHS, MPS IS: MPS IH (Hurler syndrome) patients; MPS IHS (Hurler-Scheie syndrome) patients; and MPS IS (Scheie syndrome) patients
- MPS II: Hunter syndrome patients
- MPS IV: Morquio syndrome patients who will be considered for enrollment in the study on an individual basis
- MPS VI: Maroteaux-Lamy syndrome patients
- MPS VII: Sly syndrome patients who will be considered for enrollment in the study on an individual basis

SUMMARY:
Neurobehavioral function and quality of life are compromised in many patients with mucopolysaccharidosis (MPS) disorders. The long-term goals of this research are to: 1) more accurately inform patients/parents regarding potential neurobehavioral outcomes; 2) develop sensitive measures of disease progression and central nervous system (CNS) treatment outcome; and 3) help clinical researchers develop direct treatments for specific brain structures/functions. The investigators hypothesize that specific and localized neuroimaging and neuropsychological findings and their relationship will be distinct for each MPS disorder. It is further hypothesized that without treatment, functions will decline and structure will change over time in a predictable fashion, and will be related to locus of abnormality and stage of disease.

DETAILED DESCRIPTION:
The mucopolysaccharidoses (MPS diseases) are lysosomal disorders (inborn errors of metabolism) that progressively affect most organ systems in the body, usually beginning in childhood. Recent treatment advances have produced amelioration of some of these malfunctions, but notably brain and bone have been difficult to effectively treat. This research addresses the brain abnormalities in the MPS disorders, about which little is known.

The objectives of this research are:

1. to identify abnormalities of central nervous system (CNS) structure and function as well as to measure quality-of-life (QOL) in both treated and untreated MPS patients over time. The investigators will accomplish this through longitudinal studies of enrolled patients in designated centers in North America.
2. to develop quantitative measurements of change, including direct measurement of neuropsychological function; surrogate MRI markers; and biomarkers to measure stage of disease and treatment outcomes.
3. to examine the degree to which independent variables have an impact on both functional and structural outcome. Independent variables may include, but are not limited to: age at first treatment, severity of disease, types of medical abnormalities, nature of genetic mutation, medical events, and sensory abnormalities.
4. to examine how treatments such as Enzyme Replacement Therapy (ERT), Hematopoietic Cell Transplant (HCT), substrate reduction, and other palliative and rehabilitative therapies differentially affect CNS structure and function, as well as the subject's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Any MPS I, II, IV, VI or VII child or adult aged 6 years of age or older

Exclusion Criteria:

* Exclusion Criteria for Neuroimaging:

  * Participants with:

    * Pacemakers
    * Any indwelling electronic device including programmable shunts
    * Orthodontic braces unless they are not made of metal
    * Other implanted metal in the body other than titanium
    * Unable to stay still during MRI because of low cognitive function, behavioral dysregulation, or young age, if the patient is not a clinical patient having sedation/anesthesia
    * Pregnancy
* Exclusion Criteria for Neuropsychological and Neurobehavioral Testing

  * Participants who:

    * Are too functionally impaired for testing

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is comprised of patients who have a verified diagnosis of MPS I, II, IV, VI or VII, aged 6 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Ability (IQ) | Baseline, Year 1, Year 2, Year 3
  Age-appropriate IQ tests will be administered at baseline and during subject's annual visit.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, Year 1, Year 2, Year 3
  Age-appropriate Quality of Life measures will be administered at baseline and during subject's annual visit.
Change in Neuropsychological Status | Baseline, Year 1, Year 2, Year 3
  Memory, Attention, Visual Spatial, and Visual Motor functions will be assessed with age-appropriate measures administered at baseline and during subject's annual visit.
Change in Emotional and Behavioral Health | Baseline, Year 1, Year 2, Year 3
  Age-appropriate measures of emotional and behavioral health will be administered at baseline and during subject's annual visit.
Change Shown in Magnetic Resonance Imaging of the Brain | Baseline, Year 1, Year 2, Year 3
  Magnetic resonance imaging of each subject's brain will be performed at baseline and during subject's annual visit to acquire volumetric, diffusion tensor imaging (DTI), and resting state data. These data will be analyzed to identify any changes occurring over time.
Change in Adaptive Functions | Baseline, Year 1, Year 2, Year 3
  Vineland Adaptive Behavior Scales, a measure of communication, daily living skills, socialization and motor function, will be administered at baseline and during subject's annual visit.

CONTACTS AND LOCATIONS:
Overall Officials: Chester B. Whitley, M.D., Ph.D., Principal Investigator — University of Minnesota; Ashley Schneider, Study Director — University of Minnesota; Paul Harmatz, M.D., Study Chair — Oakland Children's Hospital; Michal Inbar-Feigenberg, M.D., Study Chair — Hospital for Sick Children, Toronto, Ontario, CA; Heather Lau, M.D., Study Chair — New York University
Locations (4):
- United States (3):
  - Oakland Children's Hospital, Oakland, California
  - University of Minnesota, Minneapolis, Minnesota
  - New York University, New York, New York
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study's data will be input to the Data Management and Coordinating Center ("DMCC"), which is a part of the NIH-funded Rare Diseases Clinical Research Network. Eventually the data will be available to researchers on the database of Genotypes and Phenotypes ("dbGaP"), a part of National Center for Biotechnology Information, U.S. National Library of Medicine.

REFERENCES:
- [Background] Aldenhoven M, Wynn RF, Orchard PJ, O'Meara A, Veys P, Fischer A, Valayannopoulos V, Neven B, Rovelli A, Prasad VK, Tolar J, Allewelt H, Jones SA, Parini R, Renard M, Bordon V, Wulffraat NM, de Koning TJ, Shapiro EG, Kurtzberg J, Boelens JJ. Long-term outcome of Hurler syndrome patients after hematopoietic cell transplantation: an international multicenter study. Blood. 2015 Mar 26;125(13):2164-72. doi: 10.1182/blood-2014-11-608075. Epub 2015 Jan 26. PMID 25624320
- [Background] Braunlin E, Orchard PJ, Whitley CB, Schroeder L, Reed RC, Manivel JC. Unexpected coronary artery findings in mucopolysaccharidosis. Report of four cases and literature review. Cardiovasc Pathol. 2014 May-Jun;23(3):145-51. doi: 10.1016/j.carpath.2014.01.001. Epub 2014 Jan 10. PMID 24508139
- [Background] Stevenson DA, Rudser K, Kunin-Batson A, Fung EB, Viskochil D, Shapiro E, Orchard PJ, Whitley CB, Polgreen LE. Biomarkers of bone remodeling in children with mucopolysaccharidosis types I, II, and VI. J Pediatr Rehabil Med. 2014;7(2):159-65. doi: 10.3233/PRM-140285. PMID 25096868
- [Background] Polgreen LE, Thomas W, Orchard PJ, Whitley CB, Miller BS. Effect of recombinant human growth hormone on changes in height, bone mineral density, and body composition over 1-2 years in children with Hurler or Hunter syndrome. Mol Genet Metab. 2014 Feb;111(2):101-6. doi: 10.1016/j.ymgme.2013.11.013. Epub 2013 Dec 11. PMID 24368158
- [Background] Taylor NE, Dengel DR, Lund TC, Rudser KD, Orchard PJ, Steinberger J, Whitley CB, Polgreen LE. Isokinetic muscle strength differences in patients with mucopolysaccharidosis I, II, and VI. J Pediatr Rehabil Med. 2014;7(4):353-60. doi: 10.3233/PRM-140305. PMID 25547887
- [Background] Wolf DA, Banerjee S, Hackett PB, Whitley CB, McIvor RS, Low WC. Gene therapy for neurologic manifestations of mucopolysaccharidoses. Expert Opin Drug Deliv. 2015 Feb;12(2):283-96. doi: 10.1517/17425247.2015.966682. Epub 2014 Dec 16. PMID 25510418
- [Background] Ou L, Herzog TL, Wilmot CM, Whitley CB. Standardization of alpha-L-iduronidase enzyme assay with Michaelis-Menten kinetics. Mol Genet Metab. 2014 Feb;111(2):113-5. doi: 10.1016/j.ymgme.2013.11.009. Epub 2013 Nov 26. PMID 24332804
- [Background] Kunin-Batson AS, Shapiro EG, Rudser KD, Lavery CA, Bjoraker KJ, Jones SA, Wynn RF, Vellodi A, Tolar J, Orchard PJ, Wraith JE. Long-Term Cognitive and Functional Outcomes in Children with Mucopolysaccharidosis (MPS)-IH (Hurler Syndrome) Treated with Hematopoietic Cell Transplantation. JIMD Rep. 2016;29:95-102. doi: 10.1007/8904_2015_521. Epub 2016 Jan 30. PMID 26825088
- [Background] Polgreen LE, Kunin-Batson A, Rudser K, Vehe RK, Utz JJ, Whitley CB, Dickson P. Pilot study of the safety and effect of adalimumab on pain, physical function, and musculoskeletal disease in mucopolysaccharidosis types I and II. Mol Genet Metab Rep. 2017 Jan 15;10:75-80. doi: 10.1016/j.ymgmr.2017.01.002. eCollection 2017 Mar. PMID 28119823
- [Background] Eisengart JB, Rudser KD, Xue Y, Orchard P, Miller W, Lund T, Van der Ploeg A, Mercer J, Jones S, Mengel KE, Gokce S, Guffon N, Giugliani R, de Souza CFM, Shapiro EG, Whitley CB. Long-term outcomes of systemic therapies for Hurler syndrome: an international multicenter comparison. Genet Med. 2018 Nov;20(11):1423-1429. doi: 10.1038/gim.2018.29. Epub 2018 Mar 8. PMID 29517765
- [Background] Janzen D, Delaney KA, Shapiro EG. Cognitive and adaptive measurement endpoints for clinical trials in mucopolysaccharidoses types I, II, and III: A review of the literature. Mol Genet Metab. 2017 Jun;121(2):57-69. doi: 10.1016/j.ymgme.2017.05.005. Epub 2017 May 8. PMID 28506702
- [Background] van der Lee JH, Morton J, Adams HR, Clarke L, Ebbink BJ, Escolar ML, Giugliani R, Harmatz P, Hogan M, Jones S, Kearney S, Muenzer J, Rust S, Semrud-Clikeman M, Wijburg FA, Yu ZF, Janzen D, Shapiro E. Cognitive endpoints for therapy development for neuronopathic mucopolysaccharidoses: Results of a consensus procedure. Mol Genet Metab. 2017 Jun;121(2):70-79. doi: 10.1016/j.ymgme.2017.05.004. Epub 2017 May 6. PMID 28501294
- [Background] Nestrasil I, Vedolin L. Quantitative neuroimaging in mucopolysaccharidoses clinical trials. Mol Genet Metab. 2017 Dec;122S:17-24. doi: 10.1016/j.ymgme.2017.09.006. Epub 2017 Sep 15. PMID 29111092
- [Background] Whitley CB, Cleary M, Eugen Mengel K, Harmatz P, Shapiro E, Nestrasil I, Haslett P, Whiteman D, Alexanderian D. Observational Prospective Natural History of Patients with Sanfilippo Syndrome Type B. J Pediatr. 2018 Jun;197:198-206.e2. doi: 10.1016/j.jpeds.2018.01.044. Epub 2018 Apr 13. PMID 29661560
- [Result] Shapiro E, Guler OE, Rudser K, Delaney K, Bjoraker K, Whitley C, Tolar J, Orchard P, Provenzale J, Thomas KM. An exploratory study of brain function and structure in mucopolysaccharidosis type I: long term observations following hematopoietic cell transplantation (HCT). Mol Genet Metab. 2012 Sep;107(1-2):116-21. doi: 10.1016/j.ymgme.2012.07.016. Epub 2012 Jul 20. PMID 22867884
- [Result] Eisengart JB, Rudser KD, Tolar J, Orchard PJ, Kivisto T, Ziegler RS, Whitley CB, Shapiro EG. Enzyme replacement is associated with better cognitive outcomes after transplant in Hurler syndrome. J Pediatr. 2013 Feb;162(2):375-80.e1. doi: 10.1016/j.jpeds.2012.07.052. Epub 2012 Sep 10. PMID 22974573
- [Result] Shapiro EG, Nestrasil I, Rudser K, Delaney K, Kovac V, Ahmed A, Yund B, Orchard PJ, Eisengart J, Niklason GR, Raiman J, Mamak E, Cowan MJ, Bailey-Olson M, Harmatz P, Shankar SP, Cagle S, Ali N, Steiner RD, Wozniak J, Lim KO, Whitley CB. Neurocognition across the spectrum of mucopolysaccharidosis type I: Age, severity, and treatment. Mol Genet Metab. 2015 Sep-Oct;116(1-2):61-8. doi: 10.1016/j.ymgme.2015.06.002. Epub 2015 Jun 17. PMID 26095521
- [Result] Yund B, Rudser K, Ahmed A, Kovac V, Nestrasil I, Raiman J, Mamak E, Harmatz P, Steiner R, Lau H, Vekaria P, Wozniak JR, Lim KO, Delaney K, Whitley C, Shapiro EG. Cognitive, medical, and neuroimaging characteristics of attenuated mucopolysaccharidosis type II. Mol Genet Metab. 2015 Feb;114(2):170-7. doi: 10.1016/j.ymgme.2014.12.299. Epub 2014 Dec 9. PMID 25541100
- [Result] Ahmed A, Whitley CB, Cooksley R, Rudser K, Cagle S, Ali N, Delaney K, Yund B, Shapiro E. Neurocognitive and neuropsychiatric phenotypes associated with the mutation L238Q of the alpha-L-iduronidase gene in Hurler-Scheie syndrome. Mol Genet Metab. 2014 Feb;111(2):123-7. doi: 10.1016/j.ymgme.2013.11.014. Epub 2013 Dec 12. PMID 24368159
- [Result] Shapiro EG, Rudser K, Ahmed A, Steiner RD, Delaney KA, Yund B, King K, Kunin-Batson A, Eisengart J, Whitley CB. A longitudinal study of emotional adjustment, quality of life and adaptive function in attenuated MPS II. Mol Genet Metab Rep. 2016 Apr 1;7:32-9. doi: 10.1016/j.ymgmr.2016.03.005. eCollection 2016 Jun. PMID 27114914
- [Result] Ahmed A, Shapiro E, Rudser K, Kunin-Batson A, King K, Whitley CB. Association of somatic burden of disease with age and neuropsychological measures in attenuated mucopolysaccharidosis types I, II and VI. Mol Genet Metab Rep. 2016 Apr 1;7:27-31. doi: 10.1016/j.ymgmr.2016.03.006. eCollection 2016 Jun. PMID 27114913
- [Result] Ahmed A, Rudser K, Kunin-Batson A, Delaney K, Whitley C, Shapiro E. Mucopolysaccharidosis (MPS) Physical Symptom Score: Development, Reliability, and Validity. JIMD Rep. 2016;26:61-8. doi: 10.1007/8904_2015_485. Epub 2015 Aug 25. PMID 26303610
- [Result] Polgreen LE, Vehe RK, Rudser K, Kunin-Batson A, Utz JJ, Dickson P, Shapiro E, Whitley CB. Elevated TNF-alpha is associated with pain and physical disability in mucopolysaccharidosis types I, II, and VI. Mol Genet Metab. 2016 Apr;117(4):427-30. doi: 10.1016/j.ymgme.2016.01.012. Epub 2016 Jan 28. PMID 26873528
- [Result] Eisengart JB, Jarnes J, Ahmed A, Nestrasil I, Ziegler R, Delaney K, Shapiro E, Whitley C. Long-term cognitive and somatic outcomes of enzyme replacement therapy in untransplanted Hurler syndrome. Mol Genet Metab Rep. 2017 Sep 27;13:64-68. doi: 10.1016/j.ymgmr.2017.07.012. eCollection 2017 Dec. PMID 28983455
- [Result] Shapiro EG, Whitley CB, Eisengart JB. Beneath the floor: re-analysis of neurodevelopmental outcomes in untreated Hurler syndrome. Orphanet J Rare Dis. 2018 May 11;13(1):76. doi: 10.1186/s13023-018-0817-3. PMID 29751845
- [Derived] Kovac V, Shapiro EG, Rudser KD, Mueller BA, Eisengart JB, Delaney KA, Ahmed A, King KE, Yund BD, Cowan MJ, Raiman J, Mamak EG, Harmatz PR, Shankar SP, Ali N, Cagle SR, Wozniak JR, Lim KO, Orchard PJ, Whitley CB, Nestrasil I. Quantitative brain MRI morphology in severe and attenuated forms of mucopolysaccharidosis type I. Mol Genet Metab. 2022 Feb;135(2):122-132. doi: 10.1016/j.ymgme.2022.01.001. Epub 2022 Jan 7. PMID 35012890
- See also: The National MPS Society (in the United States) — http://mpssociety.org/
- See also: The Canadian MPS Society's own site — https://www.mpssociety.ca/